CLINICAL TRIAL: NCT01456546
Title: Impact of CYP2C19*17 on the Pharmacokinetics of Proguanil and Clopidogrel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Rasmus Steen Pedersen, Assistant Professor, University of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AKF-380
Record Dates: First submitted 2011-10-06; First posted 2011-10-20 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: CYP2C19 Genotypes
Keywords: CYP2C19*17; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Proguanil; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Period A: proguanil (Active Comparator): Proguanil pharmacokinetics
  Interventions: Drug: Proguanil
- Period B: clopidogrel (Active Comparator): Clopidogrel pharmacokinetics
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Proguanil — 2x350 mg Malarone followed by 3 days of blood- and urine sampling
  Arms: Period A: proguanil
Drug: Clopidogrel — 2x300 mg Plavix followed by 7 hours days of blood sampling
  Arms: Period B: clopidogrel

SUMMARY:
The aim of this study is to investigate if the genetic variant CYP2C19*17 affects the pharmacokinetics of proguanil and clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Written consent
* Age 18-65
* CYP2C19*1 and or CYP2C19*17 genotype.

Exclusion Criteria:

* Daily medication
* Alcohol abuse
* Pregnancy
* Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Proguanil pharmacokinetics. Primary endpoint is cycloguanil formation clearance. | Hours after administration: 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 10, 24, 31, 48, 55
  Based on blood- and urine-concentrations of proguanil and the metabolites cycloguanil and 4-chlorphenylbiguanid a comparison of the pharmacokinetic parameters (AUC, Cmax, Tmax, T1/2) between the three groups of genotypes (CYP2C19*1/*1, CYP2C19*1/*17 and CYP2C19*17/*17) will be made.

SECONDARY OUTCOMES:
Pharmacokinetics of the derivatised active clopidogrel metabolite. | Hours after administration: 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7
  Based on blood-concentrations of the derivatised active metabolite of clopidogrel a comparison of the pharmacokinetic parameters (AUC, Cmax, Tmax, T1/2) between the three groups of genotypes (CYP2C19*1/*1, CYP2C19*1/*17 and CYP2C19*17/*17) will be made.
  Secondly, a comparison of the platelet inhibitory of clopidogrel between the three groups of genotypes (CYP2C19*1/*1, CYP2C19*1/*17 and CYP2C19*17/*17) will be made using the VerifyNow® P2Y12 Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology, University of Southern Denmark, Odense, Fyn, Denmark